CLINICAL TRIAL: NCT06550752
Title: Intracavernous Injection of Umbilical Cord Stem Cells and Platelet-Rich Plasma for the Treatment of Erectile Dysfunction
Brief Title: Erectile Dysfunction Treatment Using Stem Cells
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: COR clinic of Regenerative Medicine (Network)
Responsible Party: Principal Investigator, Nada Alaaeddine, Dean of health Sciences at MUBS, Modern University for Business and Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2024-cor002
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mixture UC-MSCs and PRP (Experimental): A mixture of UCSCs and PRP will be injected into the corpora cavernosa of the penis of each patient. The injection will be done at four points along the shaft on both sides of the penis. The injection procedure will be performed once per month for a total duration of three months. Each patient received a dosage of 10 million cells per injection session.
  Interventions: Combination Product: UC-MSCs and PRP

INTERVENTIONS:
Combination Product: UC-MSCs and PRP — UC-MSCs are progenitor cells that can differentiate into various types of cells in the body and have the ability to regenerate and repair damaged tissue. During repair and regeneration, these cells secrete expedient and powerful bioactive paracrine factors including cytokines, chemokines, collagen, fibronectin, and growth factors promoting tissue repair, angiogenesis, and the regeneration of nerve cells as well as regulating cellular pathways including immunomodulation and inflammatory responses. Additionally, PRP contains numerous growth factors and cytokines, including vascular endothelial growth factor (VEGF), transforming growth factor beta-1 and beta-2 (TGF-β1/2), platelet-derived growth factor (PDGF), insulin-like growth factor (IGF), interleukin 8 and matrix metalloproteinases 2,9. The combined effect of these factors provided by PRP injections is proposed to have anti- inflammatory, reparative, neuroprotective and neurotrophic effects that contribute to the treatment of ED.

SUMMARY:
A prospective clinical study to investigate the safety and efficacy of intracavernosal injections of umbilical cord stem cells (UCSCs) combined with platelet-rich plasma (PRP) for erectile dysfunction

DETAILED DESCRIPTION:
Umbilical cord mesenchymal stem cells (UC-MSCs) combined with platelet-rich plasma (PRP) will be injected into the corpora cavernosa of the penis of male patients with erectile dysfunction. The injection will be done at four points along the shaft on both sides of the penis. Penile Doppler ultrasonography will be performed on all patients before the initiation of the treatment. This assessment will be conducted to establish a baseline measurement of penile blood flow in both left and right sides of the penis. Subsequently, after four months of treatment, penile duplex Doppler ultrasonography will be repeated to compare the penile doppler before and after treatment. Statistical analyses will be performed using IBM SPSS Statistics for Windows, version 26.

ELIGIBILITY:
Inclusion Criteria:

* male patient with erectile dysfunction

Exclusion Criteria:

* undergo other treatments for erectile dysfunction

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — this trial studies the erectile dysfunction in male patients
Enrollment: 30 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Penile Doppler ultrasonography for assessment of erectile function | before treatment and after 4 months
  Penile Doppler ultrasonography will be used to evaluate erectile function by measuring peak systolic velocity (PSV) in the penile arteries. This parameter will be assessed before the initiation of the treatment and after 4 months of treatment to evaluate blood flow in the penile arteries. The primary outcome will focus on changes in PSV, which will be compared between the baseline and post-treatment assessments to determine the efficacy of the intervention.

SECONDARY OUTCOMES:
Adverse effects | Directly after the injection and after two weeks
  patients will be asked to report any adverse effects related to the injected product or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nada Alaaeddine, PhD, Principal Investigator — COR clinic for Regenerative Medicine
Locations (1):
- COR clinic for Regenerative Medicine, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No